CLINICAL TRIAL: NCT02934334
Title: A Collaborative Investigation of Predictors of Relapse in Major Depressive Disorder: CAN-BIND-1 Extension Study
Brief Title: Wellness Monitoring for Major Depressive Disorder
Acronym: CBN-Well
Status: Completed | Type: Observational
Sponsor: Sidney Kennedy (Other)
Responsible Party: Sponsor-Investigator, Sidney Kennedy, Senior Scientist, Psychiatrist, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Other Study IDs: REB 15-9780-AE
Record Dates: First submitted 2016-10-12; First posted 2016-10-14 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Major Depressive Disorder
Keywords: major depression; major depressive episode; biomarkers; relapse; near term relapse; m-health
MeSH Terms: conditions — Depressive Disorder, Major; Recurrence | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At each 8 week visit, blood samples for biochemical, genomic, and proteomic analysis will be collected and stored at -80'C freezer.
  Plasma: Venous blood will be collected in 6mL and 10ml EDTA blood tubes, followed by centrifugation in a refrigerated centrifuge to obtain the plasma. Two milliliters of plasma from each tube will be divided into 8 cryovials (500µL).
  DNA for methylation analysis: Venous blood will be collected in 8.5 mL PAXgene DNA tubes.
  DNA for studying histone modifications: Venous blood will be collected in 6mL EDTA blood tubes and the mixed contents will be divided evenly into three 2 mL screw-cap tubes.
  RNA for mRNA and miRNA sequencing: Venous blood will be collected in 6mL EDTA blood tubes and the mixed contents will be passed through LeukoLOCK filters according to the manufacturer's instructions.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- MDD: Major Depressive Disorder
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational

SUMMARY:
The Wellness Monitoring for Major Depressive Disorder (MDD) study is a prospective, longitudinal, observational study aimed at identifying biomarkers of relapse in MDD. Results may help refine clinical approach to relapse management, and may ultimately help MDD patients sustain wellness while on antidepressant medication.

DETAILED DESCRIPTION:
This study involves a naturalistic follow up of responders from the study entitled "Integrated biological markers for the prediction of treatment response in depression", or the CAN-BIND-1 study. In addition, this study is also open to other participants who completed other CAN-BIND studies, as well as remitters who meet the inclusion criteria. Since patients usually seek medical attention only after relapse has occurred, imminent precursors to relapse are not well known. In this study, participants who are currently responding to an oral antidepressant treatment regimen and/or therapeutic intervention will be monitored over a minimum period of 13 months, which provides a unique opportunity to discover near-term biomarkers of relapse.

The study is conducted in partnership with Janssen Research & Development and utilizes remote monitoring technology for data gathering.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-V criteria for Major Depressive Episode (MDE) in MDD as determined by MINI.
* MADRS total score of equal to or less than 14.
* In the current MDE, patient must currently be responding to an antidepressant medication or a combination of treatments for MDD.
* Willing and able to complete self-reported assessments via a study-specific smartphone (LogPad), including sufficient fluency in English.
* Willing to wear GT9X Link, a wrist-worn device for the duration of the study.

Exclusion Criteria:

* Axis I diagnosis, other than MDD, that is considered the primary diagnosis.
* Bipolar I or Bipolar II diagnosis (lifetime), MDD with psychotic features (lifetime), schizophrenia, or schizoaffective disorder.
* Presence of a significant Axis II diagnosis (borderline, antisocial).
* High suicidal risk, defined by clinician judgement.
* History of drug or alcohol use, with severity of at least moderate or severe, according to DSM criteria, within 6 months before screening.
* Presence of significant neurological disorders, head trauma, or other unstable medical conditions.
* Received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 90 days before screening or is currently enrolled in an investigational study.
* Has a condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (e.g. compromise well being) or that could prevent, limit, or confound the protocol-specified assessments.
* Subject is an employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, or is a family member of an employee or the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women between 18 to 65 years of age who have previously met DSM-V criteria for Major Depressive Episode (MDE) in MDD as determined by MINI, (1) who participated in CAN-BIND-1 protocol, (2) other CAN-BIND studies, and (3) other remitters who meet the inclusion criteria who are currently responding to antidepressant medication or a combination of treatments.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-02-25 (Actual)

PRIMARY OUTCOMES:
Rate of MDD Patients with Near Term Relapse | Baseline up to the one year enrolment period for the last-subject-in.
  Relapse is defined as:
  1. MADRS total score equal to or greater than 22 on at least 2 consecutive visits (scheduled or unscheduled);
  2. Hospitalization for worsening of depression;
  3. Suicidal ideation with intent, or suicidal behaviour;
  4. Others. Investigators will be asked to describe.

CONTACTS AND LOCATIONS:
Overall Officials: Sidney H. Kennedy, MD, Principal Investigator — University Health Network, Toronto
Locations (5):
- Canada (5):
  - University of Calgary, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - McMaster University, Hamilton, Ontario
  - Queen's University, Kingston, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
This study is funded in part by the Ontario Brain Institute (OBI). Data collected from this study is entered into a research database called "Brain-CODE", deployed at a High Performance Computer Virtual Lab (HPCVL). The HPCVL supports the regulatory-compliant (e.g., 21 CRF Part 11, HIPAA, PIPEDA) processes for securing privacy of healthcare data.

REFERENCES:
- [Background] Kennedy SH, Downar J, Evans KR, Feilotter H, Lam RW, MacQueen GM, Milev R, Parikh SV, Rotzinger S, Soares C. The Canadian Biomarker Integration Network in Depression (CAN-BIND): advances in response prediction. Curr Pharm Des. 2012;18(36):5976-89. doi: 10.2174/138161212803523635. PMID 22681173
- [Background] Lam RW, Milev R, Rotzinger S, Andreazza AC, Blier P, Brenner C, Daskalakis ZJ, Dharsee M, Downar J, Evans KR, Farzan F, Foster JA, Frey BN, Geraci J, Giacobbe P, Feilotter HE, Hall GB, Harkness KL, Hassel S, Ismail Z, Leri F, Liotti M, MacQueen GM, McAndrews MP, Minuzzi L, Muller DJ, Parikh SV, Placenza FM, Quilty LC, Ravindran AV, Salomons TV, Soares CN, Strother SC, Turecki G, Vaccarino AL, Vila-Rodriguez F, Kennedy SH; CAN-BIND Investigator Team. Discovering biomarkers for antidepressant response: protocol from the Canadian biomarker integration network in depression (CAN-BIND) and clinical characteristics of the first patient cohort. BMC Psychiatry. 2016 Apr 16;16:105. doi: 10.1186/s12888-016-0785-x. PMID 27084692
- [Background] Vaccarino AL, Evans KR, Kalali AH, Kennedy SH, Engelhardt N, Frey BN, Greist JH, Kobak KA, Lam RW, MacQueen G, Milev R, Placenza FM, Ravindran AV, Sheehan DV, Sills T, Williams JB. The Depression Inventory Development Workgroup: A Collaborative, Empirically Driven Initiative to Develop a New Assessment Tool for Major Depressive Disorder. Innov Clin Neurosci. 2016 Oct 1;13(9-10):20-31. eCollection 2016 Sep-Oct. PMID 27974997
- See also: Press release — http://www.newswire.ca/news-releases/new-collaboration-established-to-tackle-depression-relapse-with-mobile-technology-587452871.html